CLINICAL TRIAL: NCT03186417
Title: Cell-Based Therapy in Rheumatoid Arthritis: Proof of Concept Phase 1 Trial
Brief Title: Mesenchymal Stem Cells in Early Rheumatoid Arthritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow enrollment during covid and lack of funds to continue
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Nora G. Singer, Physician, MetroHealth Medical Center
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB16-00587; R21AR069226 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis, Rheumatoid, Stem Cells, Mesenchymal, Autoimmune
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Intervention Model Description: This is a dose escalation study using three groups (or cohorts) of patients randomly assigned within treatment groups to MSCs or placebo. The first group will consist of 5 patients who receive MSCs and one patient who receives placebo, the second and third group will consist of five patients each who receive MSCs and two patients who receive placebo. The three doses are 2 million hMSCs/kg (Cohort 1), 4 million hMSCs/kg (Cohort 2), and 6 million hMSCs/kg (Cohort 3) and placebo control of normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 2 million human MSC (hMSC)/kg infusion versus placebo infusion
  Interventions: Biological: 2 million hMSC/kg; Biological: placebo
- Cohort 2 (Experimental): 4 million hMSC/kg infusion versus placebo infusion
  Interventions: Biological: 4 million hMSC/kg; Biological: placebo
- Cohort 3 (Experimental): 6 million hMSC/kg infusion versus placebo infusion
  Interventions: Biological: 6 million hMSC/kg; Biological: placebo

INTERVENTIONS:
Biological: 2 million hMSC/kg — 2 million hMSCs/kg infusion
  Arms: Cohort 1
Biological: 4 million hMSC/kg — 4 million hMSC/kg infusion
  Arms: Cohort 2
Biological: 6 million hMSC/kg — 6 million hMSC/kg infusion
  Arms: Cohort 3
Biological: placebo — placebo infusion

SUMMARY:
This is a prospective, multicenter, double-blind, placebo controlled interventional study to evaluate the safety and efficacy of allogeneic mesenchymal stem cells (MSCs) in 20 patients with new onset Rheumatoid Arthritis (RA). The study is a single dose, phase I clinical trial and is the first time that this product will be infused in RA patients. The study duration is approximately fourteen months from time of screening to completion.

Research hypothesis: The investigators hypothesize that when administered therapeutically, MSCs will induce healthy immune responses and will reduce RA disease activity. This study is primarily focused on demonstrating the safety of this approach.

DETAILED DESCRIPTION:
This is a prospective, multicenter (with two performance sites under the auspices of Case Western Reserve University Clinical and Translational Science Award (CWRU CTSA) at University Hospitals and at MetroHealth Medical Center), double-blind, placebo-controlled, interventional study to evaluate the safety and efficacy of allogeneic mesenchymal stem cells (MSCs) infusion in 20 new onset Rheumatoid Arthritis (RA) patients with moderate to high disease activity despite adequate doses of methotrexate (MTX) for 12 weeks (at least 10 weeks of which has been at a dose of >/=15 mg per week). The study is a single dose, phase I clinical trial, and this is the first time that this product will be infused in RA patients. After a screening period, the baseline visit will be conducted. Patients will halt their concomitant MTX 3 days prior to the MSC infusion and may resume their methotrexate at Day 7 following MSC infusion based on their disease activity score. This is a dose escalation study of a total of 20 patients with three groups of five patients each and five placebo patients. Patients will be randomized to receive MSC or placebo infusion using a computer-generated randomization scheme that takes into account that there are two sites. The first cohort will consist of a total of six patients. Of these six patients, five patients each will receive a single infusion of 2 million/kg MSCs and one patient will receive placebo infusion. The second cohort will include a total of seven patients, of these seven patients; five patients will receive 4 million/kg MSCs and two patients who will receive placebo infusion. The final cohort consists of a total of seven patients. Of these seven patients, five patients will receive 6 million/kg allogeneic MSCs and two patients will receive placebo infusion. Infusion will occur on Day 0. Post-infusion study visits will occur on Days 1 (Visit 3), 7 (Visit 4), 14 (Visit 5), 28 (Visit 6), 56 (Visit 7), and weeks 24 (Visit 8), 39 (Visit 9) and 52 (Visit 10). Phone calls will occur on Day 4, 21, and 72. Subject safety and tolerability of the single dose of MSCs will be evaluated at these study visits by reviewing interval histories, administering patient questionnaires (legacy [Routine Assessment of Patient Index Data 3 (RAPID 3) / Short Form 36 (SF36)] and Patient Reported Outcome Measurement Information System (PROMIS) computer adaptive technology CAT), performing physical exams and spirometry, and obtaining safety laboratories. Special attention will be given to exacerbation of RA or "flare". This study will also explore the efficacy measures: Disease Activity Score 28-C-Reactive Protein (DAS28-CRP) and American College of Rheumatology20/50/70 (ACR20/50/70 will be calculated. Since the primary hypothesis is that infusion of MSCs will induce a state of immune tolerance, various assays to detect post-infusion changes in cells subsets, function or protein biomarker will be repeated at Day 7 and/or 14 and compared to baseline values (with-in subject comparison). Biomarkers to look at cell-subsets will be drawn. Selected patient samples will be stored for exploratory studies using Mass Cytometry (Cytof 2). Lastly, for those subjects who are agreeable to undergo the procedure, a bone marrow aspiration will be performed prior to infusion with allogeneic MSCs. MSCs from RA bone marrow will be expanded, banked, and used for future translational studies.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Recent onset rheumatoid arthritis and have known doctor diagnosis ≤ 2 years and symptoms for ≤ 2 years.
* Patients must have detectable serum auto-antibodies against cyclic citrullinated peptides and/or high titer serum rheumatoid factor at screening or prior to screening.
* Subjects must have active synovitis of at least one joint.
* Patients who have been intolerant or had inadequate response to at least twelve weeks total of methotrexate, ten weeks of which methotrexate must have been dosed at ≥15 mg per week or with low dose steroids (< 10 mg prednisone per day).
* Clinically stable with no significant changes in health status within 2 weeks prior to randomization

Exclusion Criteria:

* Prior use of DMARDs other than non-steroidals, low dose prednisone, hydroxychloroquine and methotrexate
* Use of leflunomide or sulfasalazine for more than 3 days and less than 3 half lives have passed since discontinuing. For leflunomide, wash out is permissible.
* Prior use of Biologic DMARDs
* Presence of active infection
* History of chronic viral infections including Hepatitis B or C or HIV. Treated Hepatitis C is allowed if the viral in non-detectable
* Known chronic liver disease
* Pregnant, breastfeeding, or desire to become pregnant or unwilling to practice birth control during participation in the study and for twelve months after completing the study infusion, unless surgically sterilized or postmenopausal during the study.
* Active tuberculosis (TB) requiring treatment within 3 years prior to baseline
* Latent TB diagnosed during screening that has not been appropriately treated
* History of Cancer requiring chemotherapy within the past 5 years except Human Papillomavirus (HPV) related cervical changes that are not carcinoma in situ.
* Chronic obstructive pulmonary disease or known lung disease except for mild asthma treated with bronchodilators.
* Use of an investigational agent within the 4-week period prior to screen
* If Dimethyl sulfoxide (DMSO) is used in the preparation of MSCs then subjects with known sensitivity to DMSO will be excluded
* History of Transient Ischemic Attack
* History of Cerebrovascular Accident (stroke), unless there has been no CVA for > or = 1 year after the resolution of the underlying cause of the CVA
* Clinically significant heart disease (New York Heart Association, class III and class IV).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Safety assessed by dose limiting toxicity (DLT) | 14 days following infusion
  • In addition, a DLT will be assigned if through 14 days after the infusion any grade 3-4 adverse event for pulmonary, cardiac, renal, oral mucosal or hepatic, and grade 4 adverse events for other organs occurred per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Safety assessed by dose limiting toxicity | 48 hours following infusion
  • A DLT is triggered by occurrence through 48 hours after infusion of grade ≥2 infusion-related allergic toxicities, which include rash, flushing, urticaria, dyspnea, fever ≥38°C (≥100.4°F) as scored according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse events (CTCAE) version 4.03.
Safety assessed by change in spirometry | 30 minutes following infusion
  • Changes in spirometry following infusion compared to baseline
Safety assessed by all adverse events | 52 weeks following infusion
  • Incidence and severity of adverse events

SECONDARY OUTCOMES:
Change in patient reported outcomes | Up to day 28 after infusion
  2. Change in patient reported outcomes (PROMIS CAT and legacy [RAPID 3 / SF36] -questionnaires)
DAS28-CRP | Week 52
  Changes in DAS28-CRP

CONTACTS AND LOCATIONS:
Overall Officials: Nora singer, MD, Principal Investigator — MetroHealth Medical Center
Locations (2):
- United States (2):
  - UH Hospitals Cleveland, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No